CLINICAL TRIAL: NCT00329589
Title: A Phase I Open-labeled, Dose-escalation, Safety Study of the Combination of Velcade and Chemoradiation for the Treatment of Cancer Patients
Brief Title: A Trial Using Velcade Plus Chemoradiation for Central Nervous System, Head and Neck, and Cervical Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05C.255; 2005-28 (Other: CCRRC); NCI-2009-01797 (Registry Identifier: NCI CTRP); JT 1133 (Other: JeffTrial Number)
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Brain Cancer; Head and Neck Cancer; Cervix Cancer; Central Nervous System Neoplasms
Keywords: Malignancies of the central nervous system, head and neck area; and cervix
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms; Central Nervous System Neoplasms | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CNS (Experimental): Velcade (bortezomib)
  Interventions: Drug: Velcade (bortezomib)
- Head and Neck (Experimental): Velcade (bortezomib)
  Interventions: Drug: Velcade (bortezomib)
- Cervix (Experimental): Velcade (bortezomib)
  Interventions: Drug: Velcade (bortezomib)

INTERVENTIONS:
Drug: Velcade (bortezomib)

SUMMARY:
The purpose of this study is to determine the safety of Velcade when used with chemoradiation in cancer patients.

DETAILED DESCRIPTION:
* To determine the maximum tolerated dose (MTD) and a recommended phase II dose (RP2D) of Velcade® when administered as a twice weekly 3-5 second IV bolus every 3 weeks to patients with malignancies of the brain, head and neck and cervix who receive 2-8 weeks of chemoradiation.
* To evaluate the safety and toxicity profile of Velcade® when administered on a twice weekly (days 1, 4, 8 and 11) every 3 weeks (maximum 8 weeks) concurrent with chemoradiation.
* To evaluate tumor response

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy
* Requiring at least grade 2 weeks of radiation therapy
* Solid tumors of the central nervous system, head and neck area, and cervix
* World Health Organization (WHO) performance status equal to or less than 2

Exclusion Criteria:

* Equal to or greater than grade 2 peripheral neuropathy
* Myocardial infarction within 6 months
* Hypersensitivity to bortezomib, boron, or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the safe and maximum tolerated dose of Velcade® when administered as a twice weekly 3-5 second intravenous (IV) bolus every 3 weeks to patients with malignancies of the brain, head and neck, and cervix who receive 2-8 weeks of radiotherapy | 2-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dicker, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University — http://www.kimmelcancercenter.org